CLINICAL TRIAL: NCT01419444
Title: Telemedicine Versus Traditional Treatment of Muscle Tension Dysphonia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDHMTD2011
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Muscle Tension Dysphonia
Keywords: Voice; Muscle Tension Dysphonia; Hyperfunction; Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional, Onsite Treatment (Active Comparator): Onsite treatment using airflow exercises. Patients will receive face-to-face treatment with the research speech pathologist two times per week.
  Interventions: Behavioral: Airflow Exercises for Voicing
- Telemedicine Treatment (Experimental): Participants will receive treatment via telemedicine at select AHEC sites around the state of Arkansas. Treatments will occur twice per week with the research speech pathologist.
  Interventions: Behavioral: Airflow Exercises for Voicing

INTERVENTIONS:
Behavioral: Airflow Exercises for Voicing — Gargling, Cup Bubble Blowing, and Stretch and Flow Exercises will be taught to reduce laryngeal closure and improve airflow through the glottis during voicing.

SUMMARY:
The purpose of this research is to determine whether treatment of voice disorders can be provided just as effectively using telemedicine as it can using on-site, traditional therapy. An exercise protocol for improving airflow with voicing has been demonstrated to be effective in a prior UAMS investigation (Protocol 107454). These exercises are used as part of the normal clinic routine at UAMS working with individuals with voice problems. The three exercises used are: gargling with and without voicing; cup bubble blowing with and without voicing; and, stretch and flow exercises, which involves the use of a piece of tissue to provide visual biofeedback on the ability to use proper airflow with voicing. The purpose of the exercises is to increase airflow and breathiness in the voice and reduce muscle tension. In addition, patients will be taught to use a "confidential voice" or gentle voice during speaking.

The investigators voice patients come from all over the state and many cannot return for regular treatment. Developing a way to provide treatment to them closer to home could greatly improve quality of care and quality of life. Twenty participants will participate for 12 sessions each. All participants will be evaluated at UAMS before and after treatment as part of standard care and will, upon consent, be randomized to receive treatment via telemedicine at an AHEC site or at UAMS Medical Center. Homework will be provided along with log sheets. Results of airflow measures using an airflow-recording device (Viasys, KAY/PENTAX) pre- and post treatment will determine whether telemedicine results are equal to results of traditional, on-site treatment. The investigators hypothesize that results from treatment using telemedicine will be equivalent to results for onsite, traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary or Secondary Muscle Tension Dysphonia

Exclusion Criteria:

* Head and Neck Cancer
* Spasmodic Dysphonia
* Tremor
* Respiratory Compromise
* Dysphagia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean Expiratory Airflow During Comfortable Phonation | 6 weeks
  Measured pre- and post in liters/second using Phonatory Aerodynamic System.
Voicing Efficiency | 6 weeks
  Mean Airflow during voicing efficiency task, pa-pa-pa, using Phonatory Aerodynamic System. Measured in liters/second.

SECONDARY OUTCOMES:
Voice Handicap Index Questionnaire | 6 weeks
  Patient's perceived ratings of Voice Handicap on standardized, validated questionnaire.
Consensus Auditory Perceptual Evaluation of Voice | 6 weeks
  Overall perceptual rating of voice quality made by clinician on 100 point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- UAMS Medical Center Voice and Swallowing Clinic, Little Rock, Arkansas, United States